CLINICAL TRIAL: NCT05736705
Title: Randomized Controlled Trial Comparing Outcomes of Monopolar Current Cutting Knife and Bipolar RFA Knife in Esophageal Endoscopic Submucosal Dissection
Brief Title: Monopolar and Bipolar in Esophageal ESD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study being withdrawn as it is re-written now as a prospective study. Please reference new study
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Salmaan Azam Jawaid, MD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-52921
Record Dates: First submitted 2023-02-13; First posted 2023-02-21 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Neoplasm; Esophageal Polyp; Endoscopic Submucosal Dissection; Bipolar Electocautery
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: Two groups with patients randomized into receiving either the standard of care monopolar electrocautery tool or bipolar electrocautery tool.
Who Masked: Participant
Masking Description: The patient will not know which electrocautery tool will be used in their procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Monopolar Electrocautery tool (Active Comparator): Patients randomized into this group will receive the standard of care monopolar tool for their endoscopic submucosal dissection procedure.
  Interventions: Procedure: Endoscopic Submucosal Dissection
- Bipolar Electrocautery tool (Experimental): Patients randomized into this group will receive the standard of care bipolar tool for their endoscopic submucosal dissection procedure.
  Interventions: Procedure: Endoscopic Submucosal Dissection; Device: Bipolar electrocautery knife

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Participants randomized in this arm will have the removal of their esophageal lesion utilizing the monopolar electrocautery knife.
  Other Names: ESD; Mucosal Resection
Device: Bipolar electrocautery knife — Participants randomized in this arm will have the removal of their esophageal lesion utilizing the bipolar electrocautery knife.
  Other Names: ESD; Mucosal Resection
  Arms: Bipolar Electrocautery tool

SUMMARY:
The objective of this study is to prospectively document the efficacy and clinical outcomes of Endoscopic Submucosal Dissection procedure that utilize either a novel Bipolar-Current ESD device or the standard monopolar electrocautery knife.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is a novel technique for the removal of esophageal lesions or polyps with high-risk features. ESD is minimally invasive and allows the removal of esophageal polyps without resorting to morbid surgery. The process of ESD includes marking the lesions selected for removal, followed by submucosal injection of a lifting agent, then circumferential incisions using a specialized knife followed by submucosal dissection of the entire lesion.

Traditionally, knifes utilizing monopolar current such as dual knife or hybrid knife were the preferred tools for endoscopic submucosal dissection. These knifes allows accurate dissection and excellent hemostasis. However, due to monopolar current generated heat, post coagulation syndrome can be seen in up to 8 to 40 % of patients. Post coagulation syndrome present with pain, fever and leukocytosis and requires supportive treatment with IV fluid and antibiotics. In addition, for large esophageal lesions, stricturing can occur after resection due to significant scar formation induced by large amounts of energy. Almost all patients with 60% of the esophageal circumference removed via monopolar knives, will develop an esophageal stricture at some point. These patients require serial esophageal dilations, and although easily managed, its development can be quite troublesome to the patient. Nevertheless, ESD is still the preferred modality for removal of these lesions, since it avoids the need for morbid surgery. Recently, a novel bipolar RFA knife were approved by FDA for the performance of ESD. The knife utilizes bipolar RFA current for submucosal dissection which can potentially expedite submucosal dissection and decrease the rates of post polypectomy syndrome and scar formation, by using significantly less energy. This bipolar knife may allow for removal of large esophageal lesions without causing major esophageal stricturing.

Our tertiary referral center Baylor St Luke's Medical Center is a center of excellence for ESD procedure and the investigators have previously reported our Esophageal ESD experience using the monopolar current knife. The goal of our protocol is to compare the performance of monopolar current cutting knife and bipolar RFA knife in esophageal endoscopic submucosal dissection.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old
* Patient is capable of providing informed consent
* Patient is referred for ESD procedure of an esophageal neoplastic lesion

Exclusion Criteria:

* Patient is < 18 years old
* Patient refused and/or unable to provide consent
* Patient is a pregnant woman
* Patients with lesions removed with other techniques besides ESD (i.e. cap EMR) or a modified ESD technique

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Speed of Endoscopic Submucosal Dissection | Day 1 (procedure day)
  The speed of endoscopic submucosal dissection as calculated by cm2/hour

SECONDARY OUTCOMES:
En-bloc resection achieved | Day 1 (procedure day)
  Endoscopist removal of entire tissue specimen as a whole
R0 Resection achieved | 1-3 days post-procedure
  Margins of tissue specimen deemed by pathologist as completely excised (R0)
Curative Resection achieved | 1-3 days post-procedure
  Complete removal of diseased tissue by endoscopic submucosal dissection procedure
Adverse events | 1 month, 3 months, 6 months, 12 months
  Collection of unanticipated medical occurrences within a 12 month time frame
Rate of esophageal stricturing post-procedure | 1-3 days post-procedure
  Calculated as a percentage of patients reported with stricturing with 1-3 days following procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States